CLINICAL TRIAL: NCT05148234
Title: A Phase I/II Trial of BMS-986253 in Myelodysplastic Syndromes
Brief Title: BMS-986253 in Myelodysplastic Syndromes
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Company closed the trial.
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Principal Investigator, Najla El Jurdi, Principal Investigator, National Cancer Institute (NCI)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: 10000356; 000356-C
Record Dates: First submitted 2021-12-04; First posted 2021-12-08 (Actual); Results first posted 2024-06-11 (Actual); Last update posted 2025-09-30 (Actual); Status verified 2025-09

CONDITIONS: Myelodysplastic Syndromes
Keywords: heterogenous clonal diseases neoplasms; Interleukin-8; DNA methyltransferase inhibitors; cytopenias; Allogeneic Hematopoietic Stem Cell Transplantation
MeSH Terms: conditions — Myelodysplastic Syndromes; Cytopenia | interventions — DNA; Decitabine; cedazuridine; HuMax-IL8; Interleukin-8

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Phase I Eligible Higher Risk (HR) Myelodysplastic Syndromes (MDS) Participants (Experimental): Escalating doses of Human Humax (HuMax)-interleukin 8 (IL-8) (BMS-986253) + deoxyribonucleic acid (DNA) methyltransferase inhibitors (DNMTi) for higher risk (HR) myelodysplastic syndromes (MDS) participants.
  Interventions: Drug: Deoxyribonucleic acid (DNA) methyltransferase inhibitors (DNMTi) Decitabine; Drug: Deoxyribonucleic acid (DNA) methyltransferase inhibitors (DNMTi) Cedazuridine; Drug: BMS-986253; Procedure: Bone Marrow Biopsy; Procedure: Bone Marrow Aspiration; Procedure: ECG
- Phase I Lower Risk (LR) Myelodysplastic Syndromes (MDS) Participants (Experimental): Escalating doses of Human Humax (HuMax)-interleukin 8 (IL-8) (BMS-986253) for lower risk (LR) myelodysplastic syndromes (MDS) participants.
  Interventions: Drug: BMS-986253; Procedure: Bone Marrow Biopsy; Procedure: Bone Marrow Aspiration; Procedure: ECG
- Phase II Higher Risk (HR) Myelodysplastic Syndromes (MDS) Participants (Experimental): Phase II dose of Human Humax (HuMax)-interleukin 8 (IL-8) (BMS-986253) + deoxyribonucleic acid (DNA) methyltransferase inhibitors (DNMTi) for higher risk (HR) myelodysplastic syndromes (MDS) participants.
  Interventions: Drug: Deoxyribonucleic acid (DNA) methyltransferase inhibitors (DNMTi) Decitabine; Drug: Deoxyribonucleic acid (DNA) methyltransferase inhibitors (DNMTi) Cedazuridine; Drug: BMS-986253; Procedure: Bone Marrow Biopsy; Procedure: Bone Marrow Aspiration; Procedure: ECG
- Phase II Lower Risk (LR) Myelodysplastic Syndromes (MDS) Participants (Experimental): Phase II dose of Human Humax (HuMax)-interleukin 8 (IL-8) (BMS-986253) for lower risk (LR) myelodysplastic syndromes (MDS) participants.
  Interventions: Drug: BMS-986253; Procedure: Bone Marrow Biopsy; Procedure: Bone Marrow Aspiration; Procedure: ECG

INTERVENTIONS:
Drug: Deoxyribonucleic acid (DNA) methyltransferase inhibitors (DNMTi) Decitabine — For Higher Risk (HR) Myelodysplastic Syndromes (MDS) cohort, the study drug of BMS-986253 will be given in combination with standard of care (SOC) Food and Drug Administration (FDA)-approved DNMTi by mouth (PO) decitabine and cedazuridine according to guidelines outlined in FDA product label. Standard of care (SOC) DNMTi will be administered via oral route once daily starting Day (D)2 of each treatment cycle through D6.
  Arms: Phase I Eligible Higher Risk (HR) Myelodysplastic Syndromes (MDS) Participants; Phase II Higher Risk (HR) Myelodysplastic Syndromes (MDS) Participants
Drug: Deoxyribonucleic acid (DNA) methyltransferase inhibitors (DNMTi) Cedazuridine — For Higher Risk (HR) Myelodysplastic Syndromes (MDS) cohort, the study drug of BMS-986253 will be given in combination with standard of care (SOC) Food and Drug Administration (FDA)-approved DNMTi by mouth (PO) decitabine and cedazuridine according to guidelines outlined in FDA product label. Standard of care (SOC) DNMTi will be administered via oral route once daily starting Day (D)2 of each treatment cycle through D6.
  Arms: Phase I Eligible Higher Risk (HR) Myelodysplastic Syndromes (MDS) Participants; Phase II Higher Risk (HR) Myelodysplastic Syndromes (MDS) Participants
Drug: BMS-986253 — Intravenous (IV) infusion, 200 mg/Vial (20 mg/mL) or 1000 mg/vial (100mg/mL). Abbreviated Title: Human Humax (HuMax)-interleukin 8 (IL-8) (BMS-986253) in Myelodysplastic Syndromes 34 Version Date: 9/08/2021 outlined in Food and Drug Administration (FDA) product label.
  Other Names: Human Humax (HuMax)-interleukin 8 (IL-8) (BMS-986253)
Procedure: Bone Marrow Biopsy — Bone marrow biopsy: required at screening/baseline, Phase I post cycle (C)
  1(C1Day(D)28 +/- 3 days) and Phase II post cycle 2 (C2D28 +/- 3 days) and post cycle 6 (C6D28 +/- 3days); and if needed clinically in the setting of aplasia or concern for disease progression.
Procedure: Bone Marrow Aspiration — Bone marrow aspiration: required at screening/baseline, Phase I post cycle (C)
  1(C1Day(D)28 +/- 3 days) and Phase II post cycle 2 (C2D28 +/- 3 days) and post cycle 6 (C6D28 +/- 3days); and if needed clinically in the setting of aplasia or concern for disease progression.
Procedure: ECG — 12-lead electrocardiogram (ECGs) will be performed at baseline only for safety.
  Other Names: Electrocardiogram

SUMMARY:
Background:

The myelodysplastic syndromes (MDS) are a group of bone marrow neoplasms. MDS mostly affect elderly people. The drugs used to treat MDS are not always effective, and the only curative treatment is stem cell transplant. Researchers want to see if a new drug can be used to treat MDS.

Objective:

To learn if HuMax-interleukin 8 (IL-8) BMS-986253 is a safe and effective treatment for MDS.

Eligibility:

Adults aged 18 and older with MDS.

Design:

Participants will be screened with a medical history, medication review, and physical exam. They will answer questions about how well they are able to take care of themselves. Their temperature, blood pressure, breathing rate, and heart rate will be monitored. They will have an electrocardiogram to see how well their heart is working. They will give blood and urine samples. They may have a bone marrow biopsy.

Participants will be assigned to a specific group. They will receive either BMS-986253 alone or in combination with deoxyribonucleic acid (DNA) methyltransferase inhibitors (DNMTi).

Treatment will be given in 28-day cycles. Participants will get BMS-986253 as an infusion on days 1 and 15 of each cycle. Some participants also will take oral DNMTi on days 2-6 of each cycle. They will receive treatment until their disease gets worse or they have bad side effects.

At study visits, some screening tests will be repeated. Some of the samples that are collected will be used for genetic testing.

About 30 days after treatment ends, participants will have a follow-up visit to see how they are doing. After that, follow up will occur via phone every 3-6 months until the study ends.

National Institutes of Health (NIH) will cover the costs for some travel expenses....

DETAILED DESCRIPTION:
Background:

The myelodysplastic syndromes (MDS) are a group of clonal bone marrow neoplasms characterized by ineffective hematopoiesis, cytopenia, and high risk for transformation to acute myeloid leukemia (AML).

MDS is primarily a disease of the elderly, with about 80% of participants being older than 65-years of age; with 10,000 new diagnoses per year in the United States (U.S.)

The only curative treatment for participants with MDS is allogeneic hematopoietic stem cell transplantation (HSCT) and only a small portion of participants are eligible. Depending on risk stratification, the median survival of high- and low-risk MDS participants is 1.5 to 5.9 years, respectively.

Deoxyribonucleic acid (DNA) methyltransferase inhibitors (DNMTi) are the standard of care therapy for high-risk MDS. However, less than half of participants respond to DNMTi, and even the best responses are transient and non-curative. More effective and less toxic therapies are needed.

Interleukin-8 (IL-8) is a proinflammatory chemokine from the chemokine (C-X-C motif) CXC family and a potent chemoattractant of granulocytes and related cells to the site of inflammation. IL-8 is uniquely upregulated and found at high levels in both the peripheral blood and bone marrow aspirates of MDS participants. In purified MDS/Acute myeloid leukemia (AML) long-term/short term stem cells and granulocyte-macrophage progenitor cells both IL-8 and the IL-8 receptor, CXCR2, are overexpressed.

Preclinical data showed that CXCR2 inhibition led to significantly reduce proliferation of leukemic cell lines. In addition, MDS cluster of differentiation 34 (CD34+) cell cultures treated with neutralizing anti-IL-8 showed improvement in erythroid colony formation.

BMS-986253 is a fully human Immunoglobulin G1 (IgG1) neutralizing antibody that showed a favorable safety profile in participants with advanced solid tumors.

Concomitant treatment with DNMTi and BMS-986253 may improve treatment responses in participants with MDS by attenuating chemoattraction of myeloid derived suppressor cells to the bone marrow, indirectly disinhibiting natural killer (NK)- and T-cell responses against MDS stem cells, reducing neoangiogenesis, and improving cytopenia.

Objectives:

Primary objectives:

Phase I: To determine the optimal biological dose (OBD) and recommended phase 2 dose (RP2D) of BMS-986253 with or without DNMTi (decitabine and cedazuridine) therapy in MDS participants, and to describe the safety and tolerability of BMS-986253.

Phase II: To determine overall response rate (ORR) to BMS-986253 with or without DNMTi (decitabine and cedazuridine) therapy in MDS, measured according to the proposed revised International Working Group (IWG) 2018 response criteria.

Eligibility:

Participants must have histologically or cytologically confirmed MDS according to 2016 World Health Organization (WHO) criteria and

* have higher risk (HR) MDS Revised International Prognostic Scoring System (R-IPSS >= 3.5) and received a minimum of 2 and maximum of 8 cycles of DNMTi for Phase I (and a maximum of 4 cycles for Phase 2), or
* have lower risk (LR) MDS (R-IPSS <3.5) and at least one cytopenia (for both Phases I and II).

Age >=18 years

Eastern Cooperative Oncology Group (ECOG) performance status <=2 (KPS >= 60%)

Design:

This study consists of two phases:

Phase I: safety evaluation with determination of optimal biological dose (OBD) of BMS-986253 with or without DNMTi (decitabine and cedazuridine), and

Phase II: efficacy evaluation of BMS-986253 with or without DNMTi (decitabine and cedazuridine)

In both Phase I and II, participants will be enrolled into two cohorts:

A) Higher-risk cohort (HR-MDS), including high-risk and higher intermediate-risk disease, defined as those with R-IPSS >= 3.5: treatment with BMS-986253 in combination with DNMTi (decitabine and cedazuridine)

B) Lower-risk cohort (LR-MDS), including low-risk and lower intermediate-risk disease participants, defined as those with R-IPSS <3.5: treatment with BMS-986253 given as monotherapy

For Phase I, the safety endpoint will be dose limiting-toxicity (DLT) by D28 with the objective of defining the OBD and RP2D for BMS-986253. In addition, follow up for safety will be assessed 100 days after the end of the treatment cycle. For Phase II, the primary endpoint will be overall response rate after 6 cycles, reported separately by cohort.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Participants must have histologically or cytologically confirmed myelodysplastic syndromes (MDS) according to 2016 World Health Organization (WHO) criteria
* And:

  * have higher-risk myelodysplastic syndrome (HR-MDS) Revised International Prognostic Scoring System (R-IPSS >= 3.5) and received a minimum of 2 and maximum of 8 prior cycles for phase I and 4 for phase II of deoxyribonucleic acid (DNA) methyltransferase inhibitors (DNMTi) therapy, or
  * have lower-risk myelodysplastic syndrome (LR-MDS) (R-IPSS <3.5),

    * and, at least one cytopenia:

      * granulocytes < 1.0 x 10^9/L and/or
      * hemoglobin < 110 g/L with signs/symptoms of symptomatic anemia or transfusion-dependency
      * platelets < 100 x 10^9/L
* Age >=18 years

  --Because no dosing or adverse event data are currently available on the use of HuMax-interleukin 8 (IL-8) BMS-986253 as monotherapy or in combination with DNMTi in participants <18 years of age, children are excluded from this study, but will be eligible for future pediatric trials.
* Eastern Cooperative Oncology Group (ECOG) performance status <=2 (Karnofsky >=60%).
* Life expectancy greater than 6 months.
* Participants must have adequate organ function as defined below:

  --total bilirubin <=1.5 X institutional upper limit of normal OR <=3 X institutional upper limit of normal in participants with Gilbert's syndrome (*except for participants with increased bilirubin levels attributed to intramedullary hemolysis, which will be allowable)
* Aspartate aminotransferase (AST)/Serum glutamic oxaloacetic transaminase (SGOT)/Alanine transaminase (ALT)/Serum glutamic-pyruvic transaminase (SGPT) <=3 X institutional upper limit of normal OR <=5 X institutional upper limit of normal if related to disease specific cause
* creatinine clearance (by Cockcroft-Gault) >=60 mL/min/1.73 m^2 for participants with creatinine levels above institutional normal.
* The effects of BMS-986253 on the developing human fetus are unknown. For this reason and because DNMTi as well as other therapeutic agents used in this trial are known to be teratogenic, women of child-bearing potential (WOCBP) and men must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, for the duration of study participation, and up to 6 months after study completion and last dose of DNMTi.
* Ability of subject to understand and the willingness to sign a written informed consent document.

EXCLUSION CRITERIA:

* For phase I: Participants with HR-MDS (R-IPSS >=3.5) that have not yet received or received less than 2 cycles of DNMTi therapy.
* Participants with LR-MDS (R-IPSS <3.5) with the following characteristics that have not yet received or are still deriving benefit from the following standard of care therapies:

  * Hemoglobin (Hgb) <10 g/dL, Epo level <500 mU/mL: Erythropoietin-stimulating agents (ESAs)
  * MDS with del5q: Lenalidomide
  * MDS with ringed sideroblasts (MDS-RS) with splicing factor 3b subunit 1 (SF3B1) mutation: Luspatercept
* Participants with platelet transfusion-refractory thrombocytopenia, with inability to keep platelet threshold above 10K/mcL with transfusions or those with ongoing or uncontrolled hemorrhagic complications.
* Participants with clinically significant neutropenia, absolute neutrophil count (ANC)<100, with frequent hospitalizations for infection (average >1 hospitalization per month in past 6 months)
* Participants who are receiving or have received any other investigational agents within 28 days before start of study

treatment.

* History of allergic reactions attributed to compounds of similar chemical or biologic composition to DNMTi or other agents used in study.
* Uncontrolled intercurrent illness including, but not limited to, ongoing or active infection, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, or psychiatric illness/social situations that would limit compliance with study requirements.
* Pregnant women or women presently breast-feeding their children are excluded due to unknown risks to a developing fetus or infant.
* Any significant disease that, in the opinion of the investigator, may impair the participant s tolerance of study treatment.
* Active or uncontrolled autoimmune diseases requiring treatment.
* Chronic hepatitis B or C infection, because potential immune impairment caused by these disorders may diminish the effectiveness of this immunologic therapy.
* Human immunodeficiency virus (HIV)-positive participants are ineligible because of the potential for decreased immune response.
* Presence of any other malignancy (except basal and squamous cell carcinoma of the skin, or stable chronic cancers on hormone or targeted therapy) for which participant received systemic anticancer treatment within 24 months prior to enrollment.
* Prior history of allogeneic hematopoietic stem cell transplantation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2022-11-29 (Actual); Primary Completion 2023-02-02 (Actual); Study Completion 2023-07-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Najla El Jurdi, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (1):
- National Institutes of Health Clinical Center, Bethesda, Maryland, United States

IPD SHARING:
Plan to Share IPD: Yes
All collected individual participant data (IPD) will be shared. In addition, all large-scale genomic sequencing data will be shared with subscribers to the database of Genotypes and Phenotypes (dbGaP).
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data from this study may be requested from other researchers after the completion of the primary endpoint. Genomic data are available once genomic data are uploaded per protocol Genomic Data Sharing (GDS) plan for as long as database is active.
Access Criteria: Data from this study may be requested by contacting the principal investigator (PI). Genomic data are made available via the database of Genotypes and Phenotypes (dbGaP) through requests to the data custodians.

REFERENCES:
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_000356-C.html

RESULTS

PARTICIPANT FLOW:
Groups:
- Phase I Dose Level -1: 600 mg Eligible Higher Risk (HR) Myelodysplastic Syndromes (MDS) Participants; Phase I Dose Level 1: 1200mg Eligible Higher Risk (HR) Myelodysplastic Syndromes (MDS) Participants; Phase I Dose Level 2: 2400 mg Eligible Higher Risk (HR) Myelodysplastic Syndromes (MDS) Participants; Phase I Dose Level 3: 3600 mg Eligible Higher Risk (HR) Myelodysplastic Syndromes (MDS) Participants: Escalating doses of Human Humax (HuMax)-interleukin 8 (IL-8) (BMS-986253) + deoxyribonucleic acid (DNA) methyltransferase inhibitors (DNMTi) for higher risk (HR) myelodysplastic syndromes (MDS) participants.
  Deoxyribonucleic acid (DNA) methyltransferase inhibitors (DNMTi) Decitabine: For Higher Risk (HR) Myelodysplastic Syndromes (MDS) cohort, the study drug of BMS-986253 will be given in combination with standard of care (SOC) Food and Drug Administration (FDA)-approved DNMTi by mouth (PO) decitabine and cedazuridine according to guidelines outlined in FDA product label. Standard of care (SOC) DNMTi will be administered via oral route once daily starting Day (D)2 of each treatment cycle through D6.
  Deoxyribonucleic acid (DNA) methyltransferase inhibitors (DNMTi) Cedazuridine: For Higher Risk (HR) Myelodysplastic Syndromes (MDS) cohort, the study drug of BMS-986253 will be given in combination with standard of care (SOC) Food and Drug Administration (FDA)-approved DNMTi by mouth (PO) decitabine and cedazuridine according to guidelines outlined in FDA product label. Standard of care (SOC) DNMTi will be administered via oral route once daily starting Day (D)2 of each treatment cycle through D6.
  BMS-986253: Intravenous (IV) infusion, 200 mg/Vial (20 mg/mL) or 1000 mg/vial (100mg/mL). Abbreviated Title: Human Humax (HuMax)-interleukin 8 (IL-8) (BMS-986253) in Myelodysplastic Syndromes 34 Version Date: 9/08/2021 outlined in Food and Drug Administration product label.
- Enrolled But Not Treated: Participant was enrolled but not treated.
Period: Phase I
Arm/Group | Phase I Dose Level -1: 600 mg Eligible Higher Risk (HR) Myelodysplastic Syndromes (MDS) Participants | Phase I Dose Level 1: 1200mg Eligible Higher Risk (HR) Myelodysplastic Syndromes (MDS) Participants | Phase I Dose Level 2: 2400 mg Eligible Higher Risk (HR) Myelodysplastic Syndromes (MDS) Participants | Phase I Dose Level 3: 3600 mg Eligible Higher Risk (HR) Myelodysplastic Syndromes (MDS) Participants | Phase I Lower Risk (LR) Myelodysplastic Syndromes (MDS) Participants | Phase II Higher Risk (HR) Myelodysplastic Syndromes (MDS) Participants | Phase II Lower Risk (LR) Myelodysplastic Syndromes (MDS) Participants | Enrolled But Not Treated
Started | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Ineligible | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Company closed the trial. | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 0
Period: Phase II
Arm/Group | Phase I Dose Level -1: 600 mg Eligible Higher Risk (HR) Myelodysplastic Syndromes (MDS) Participants | Phase I Dose Level 1: 1200mg Eligible Higher Risk (HR) Myelodysplastic Syndromes (MDS) Participants | Phase I Dose Level 2: 2400 mg Eligible Higher Risk (HR) Myelodysplastic Syndromes (MDS) Participants | Phase I Dose Level 3: 3600 mg Eligible Higher Risk (HR) Myelodysplastic Syndromes (MDS) Participants | Phase I Lower Risk (LR) Myelodysplastic Syndromes (MDS) Participants | Phase II Higher Risk (HR) Myelodysplastic Syndromes (MDS) Participants | Phase II Lower Risk (LR) Myelodysplastic Syndromes (MDS) Participants | Enrolled But Not Treated
Started | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Data was collected and reported for one participant enrolled but not treated.
Groups:
- Total: Total of all reporting groups
Arm/Group | Phase I Dose Level 1: 1200mg Eligible Higher Risk (HR) Myelodysplastic Syndromes (MDS) Participants | Enrolled But Not Treated | Total
Number analyzed (Participants) | 1 | 1 | 2
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 1 | 1 | 2
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 63 (0) | 44 (0) | 53.5 (13.44)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1 | 1 | 2
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 1 | 1
  Not Hispanic or Latino | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 1 | 1 | 2
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 1 | 1 | 2

OUTCOME MEASURES:

1. Primary Outcome: Phase I: Optimal Biological Dose (OBD) for Human Humax (HuMax)-Interleukin 8 (IL-8) (BMS-986253)
Description: OBD of BMS-986253 with and without deoxyribonucleic acid (DNA) methyltransferase inhibitors (DNMTi), as determined by dose limiting toxicity (DLT) occurring by cycle 1 day 28 (C1D28). DLT is defined as any of the following: any grade ≥ non-hematologic toxicity that is possibly, probably, or definitely related to study drug. Liver injury as defined by a positive Hy's Law. And adverse reaction that leads to dose reduction or withdrawal. OBD is the lowest tolerated dose level showing optimal biological activity, defined as maximal suppression of serum free IL-8 levels. The goal is to achieve IL-8 levels below the lower limit of detection of the assay in real time by Ultrasensitive immunoassay based on Quanterix Simoa technology. The lower limit of quantification = 0.86 pg/mL by Myriad-Rules Based Medicine (RBM).
Time Frame: First 28 days (C1D28) on up to 30 days.
Population: 1/2 participants were enrolled but not treated.
Measure: Number; unit: mg
Groups:
- All Participants: Phase I Dose Level 1: All participants who received at least on dose of drug.
Arm/Group | All Participants
Number analyzed (Participants) | 1
mg
  With DNMTi | NA — The DLT (dose limiting toxicity) refers to the highest dose of a drug that causes unacceptable or intolerable side effects or toxicities. Once we identify DLTs, we can identify the maximum tolerated doses. There is not enough data to determine OBD.
  Without DNMTi | NA — The DLT (dose limiting toxicity) refers to the highest dose of a drug that causes unacceptable or intolerable side effects or toxicities. Once we identify DLTs, we can identify the maximum tolerated doses. There is not enough data to determine OBD.

2. Primary Outcome: Phase I: Recommended Phase 2 Dose (RP2D) of Human Humax (HuMax)-Interleukin 8 (IL-8) (BMS-986253)
Description: RP2D of BMS-986253 with and without deoxyribonucleic acid (DNA) methyltransferase inhibitors (DNMTi), as determined by dose -limiting toxicity (DLT) occurring by cycle 1 day 28 (C1D28). RP2D is defined as the optimal biological dose expected to be safe and of potential efficacy. It serves as a starting point for further investigations in future phase 2 clinical trials. DLT is defined as any of the following: ang grade ≥ non-hematologic toxicity that is possibly, probably, or definitely related to study drug. Liver injury as defined by a positive Hy's Law. And adverse reaction that leads to dose reduction or withdrawal.
Time Frame: First 28 days (C1D28)
Population: 1/2 participants were enrolled but not treated.
Measure: Number; unit: mg
Arm/Group | All Participants
Number analyzed (Participants) | 1
mg
  With DNMTi | NA — The DLT (dose limiting toxicity) refers to the highest dose of a drug that causes unacceptable or intolerable side effects or toxicities. Once we identify DLTs, we can identify the Recommended Phase 2 Dose (RP2D). There is not enough data to determine MTD.
  Without DNMTi | NA — The DLT (dose limiting toxicity) refers to the highest dose of a drug that causes unacceptable or intolerable side effects or toxicities. Once we identify DLTs, we can identify the Recommended Phase 2 Dose (RP2D). There is not enough data to determine MTD.

3. Primary Outcome: Phase II: Overall Response Rate
Description: Overall response rate (ORR= Complete Remission (CR) + Partial Remission (PR) + [marrow CR + hematologic improvement (HI]) of Human Humax (HuMax)-interleukin 8 (IL-8) (BMS-986253) with and without deoxyribonucleic acid (DNA) methyltransferase inhibitors (DNMTi) after 6 cycles of therapy was assessed by the 2006 International Working Group response criteria for Myelodysplastic Syndromes. Complete Remission (CR) is bone marrow ≤55% myeloblasts with normal maturation of all cell lines. Persistent dysplasia will be noted. Partial Remission (PR) is all CR criteria if abnormal before treatment except bone marrow blasts decreased by ≥50% over pretreatment but still >5%. And cellularity and morphology not relevant.
Time Frame: 6 months
Population: This outcome measure was not done because the company closed the study prior to phase II.
Arm/Group | Phase I Dose Level 1: 1200mg Eligible Higher Risk (HR) Myelodysplastic Syndromes (MDS) Participants
Number analyzed (Participants) | 0

4. Primary Outcome: Phase I: Number of Grades 1-5 Serious and/or Non-serious Adverse Events Related to Human Humax (HuMax)-Interleukin 8 (IL-8) (BMS-986253) and Deoxyribonucleic Acid (DNA) Methyltransferase Inhibitors (DNMTi)
Description: Safety as measured by incidence of adverse events (AEs) and serious adverse events (SAEs), and AEs leading to discontinuation, death, and laboratory abnormalities. Adverse events were assessed by the Common Terminology Criteria for Adverse Events (CTCAE v5.0). A non-serious adverse event is any untoward medical occurrence. A serious adverse event is an adverse event or suspected adverse reaction that results in death, a life-threatening adverse drug experience, hospitalization, disruption of the ability to conduct normal life functions, congenital anomaly/birth defect or important medical events that jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the previous outcomes mentioned. Grade 1 is mild. Grade 2 is moderate. Grade 3 is severe. Grade 4 if life-threatening. Grade 5 is death related to adverse event.
Time Frame: First 28 days and follow up after the end of the treatment cycle; approximately 2 months.
Population: 1/2 participants were enrolled but not treated.
Measure: Number; unit: adverse events
Arm/Group | Phase I Dose Level 1: 1200mg Eligible Higher Risk (HR) Myelodysplastic Syndromes (MDS) Participants
Number analyzed (Participants) | 1
adverse events
  Grades 1-5 Serious related to BMS-986253 | 0
  Grades 1-5 Non-serious related to BMS-986253 | 0
  Grade 1 -2 Serious related to DNMTi | 0
  Grade 3 Serious related to DNMTi - Febrile neutropenia | 1
  Grade 3 Serious related to DNMTi - Skin infection | 1
  Grade 2 Non-serious related to DNMTi - Lymphocyte count decreased | 1
  Grade 3 Non-serious related to DNMTi - White blood cell decreased | 1

5. Primary Outcome: Phase II: Fraction of Participants With Clinical Response
Description: Clinical response was assessed by the assessed by the 2006 International Working Group response criteria for Myelodysplastic Syndromes and reported with 95% confidence interval. Complete Remission (CR) is bone marrow ≤55% myeloblasts with normal maturation of all cell lines. Persistent dysplasia will be noted. Partial Remission (PR) is all CR criteria if abnormal before treatment except bone marrow blasts decreased by ≥50% over pretreatment but still >5%. And cellularity and morphology not relevant. Stable disease is failure to achieve at least PR, but no evidence of progression for >8 weeks. Progression is less than 5% blasts: ≥50% increase in blasts to >5% blasts; 5%-10% blasts: ≥50% increase to 10% blasts; transfusion dependence. Relapse after CR or PR is at least 1 of the following: return to pre-treatment bone marrow blast percentage or decrement of ≥50% from maximum remission/response levels in granulocytes or platelets.
Time Frame: Study treatment until occurrence of disease progression, death, or unacceptable toxicity or until response assessment on Cycle 7 day 1 (C7D1), a maximum of 6 cycles
Population: This outcome measure was not done because the company closed the study prior to phase II.
Arm/Group | Phase I Dose Level 1: 1200mg Eligible Higher Risk (HR) Myelodysplastic Syndromes (MDS) Participants
Number analyzed (Participants) | 0

6. Secondary Outcome: Phase I: Area Under the Concentration Time Curve (AUC 0-24h) of Human Humax (HuMax)-Interleukin 8 (IL-8) (BMS-986253) in Myelodysplastic Syndromes (MDS) With and Without Deoxyribonucleic Acid (DNA) Methyltransferase Inhibitors (DNMTi)
Description: AUC is a measure of the serum concentration of drug BMS-986253 over time. It is used to characterize drug absorption.
Time Frame: Before infusion, within 30 minutes, start of infusion, 1, 4, 12, and 24 hours after end of infusion.
Population: Samples were stored but data were not analyzed because the manufacturer responsible for analyzing the samples terminated the study. No future data analysis will be conducted for samples stored for this terminated study.
Arm/Group | Phase I Dose Level 1: 1200mg Eligible Higher Risk (HR) Myelodysplastic Syndromes (MDS) Participants
Number analyzed (Participants) | 0

7. Secondary Outcome: Phase I: Half-life of Human Humax (HuMax)-Interleukin 8 (IL-8) (BMS-986253) With and Without Deoxyribonucleic Acid (DNA) Methyltransferase Inhibitors (DNMTi)
Description: Plasma decay half-life is the time measured for the plasma concentration of the drug to decrease by one half.
Time Frame: Before infusion, within 30 minutes, start of infusion, 1, 4, 12, and 24 hours after end of infusion.
Population: as for outcome 6
Arm/Group | Phase I Dose Level 1: 1200mg Eligible Higher Risk (HR) Myelodysplastic Syndromes (MDS) Participants
Number analyzed (Participants) | 0

8. Secondary Outcome: Phase I: Concentration of Human Humax (HuMax)-Interleukin 8 (IL-8) (BMS-986253) at Steady State With and Without Deoxyribonucleic Acid (DNA) Methyltransferase Inhibitors (DNMTi)
Description: Concentration of BMS-986253 at steady state in plasma.
Time Frame: Before infusion, within 30 minutes, start of infusion, 1, 4, 12, and 24 hours after end of infusion.
Population: as for outcome 6
Arm/Group | Phase I Dose Level 1: 1200mg Eligible Higher Risk (HR) Myelodysplastic Syndromes (MDS) Participants
Number analyzed (Participants) | 0

9. Secondary Outcome: Phase II: Number of Grades 1-5 Serious and/or Non-serious Adverse Events Related to Human Humax (HuMax)-Interleukin 8 (IL-8) (BMS-986253) and Deoxyribonucleic Acid (DNA) Methyltransferase Inhibitors (DNMTi)
Description: as for outcome 4
Time Frame: 1 year
Population: This outcome measure was not done because the company closed the study prior to phase II.
Arm/Group | Phase I Dose Level 1: 1200mg Eligible Higher Risk (HR) Myelodysplastic Syndromes (MDS) Participants
Number analyzed (Participants) | 0

10. Secondary Outcome: Phase II: Cytogenetic Response Rate
Description: Cytogenetic Response was assessed by the 2006 International Working Group response criteria for Myelodysplastic Syndromes. Cytogenetic complete response is disappearance of the chromosomal abnormality without appearance of new ones. Cytogenetic partial response is at least 50% reduction of the chromosomal abnormality.
Time Frame: as for outcome 5
Population: This outcome measure was not done because the company closed the study prior to phase II.
Arm/Group | Phase I Dose Level 1: 1200mg Eligible Higher Risk (HR) Myelodysplastic Syndromes (MDS) Participants
Number analyzed (Participants) | 0

11. Secondary Outcome: Phase II: Time to Best Response (Complete Remission (CR), Partial Remission (PR), Marrow CR + Hematologic Improvement (HI), HI)
Description: Time to best response (Complete Remission (CR), Partial Remission (PR), marrow CR + HI, HI) using the Kaplan-Meier method. Response was assessed by the 2006 International Working Group response criteria for Myelodysplastic Syndromes. Complete Remission (CR) is bone marrow ≤55% myeloblasts with normal maturation of all cell lines. Persistent dysplasia will be noted. Partial Remission (PR) is all CR criteria if abnormal before treatment except bone marrow blasts decreased by ≥50% over pretreatment but still >5%. And cellularity and morphology not relevant. Hematologic improvement (HI) is defined as: Erythroid response - at least 2 consecutive hemoglobin (hgb) measurements >1.5 g/dL for a period of minimum 8 weeks in an observation period of 16-24 weeks compared with the lowest mean of 2 hgb measurements within 16 weeks before treatment onset. Platelet response - absolute increase of 30x10^9/L for participants starting with >20x10^9/L platelets.
Time Frame: Time to best response
Population: This outcome measure was not done because the company closed the study prior to phase II.
Arm/Group | Phase I Dose Level 1: 1200mg Eligible Higher Risk (HR) Myelodysplastic Syndromes (MDS) Participants
Number analyzed (Participants) | 0

12. Secondary Outcome: Phase II: Disease Free Survival (DFS)
Description: DFS is defined as time to relapse for participants who achieve complete remission (CR) using the Kaplan-Meier method. Complete Remission (CR) is bone marrow ≤55% myeloblasts with normal maturation of all cell lines. Persistent dysplasia will be noted.
Time Frame: Until study closure
Population: This outcome measure was not done because the company closed the study prior to phase II.
Arm/Group | Phase I Dose Level 1: 1200mg Eligible Higher Risk (HR) Myelodysplastic Syndromes (MDS) Participants
Number analyzed (Participants) | 0

13. Secondary Outcome: Phase II: Progression Free Survival (PFS)
Description: PFS is defined as disease progression or death from Myelodysplastic Syndromes (MDS). Progression was assessed by the 2006 International Working Group response criteria for Myelodysplastic Syndromes using the Kaplan-Meier method and is defined as less than 5% blasts: ≥50% increase in blasts to >5% blasts; 5%-10% blasts: ≥50% increase to 10% blasts; 10%-20% blasts: ≥50% increase to >20% blasts; 20%-30% blasts: ≥50% increase to >30% blasts and any of the following: At least 50% decrement from maximum remission/response in granulocytes or platelets, reduction in Hgb by ≥2 g/dL, and transfusion dependence.
Time Frame: Until study closure
Population: This outcome measure was not done because the company closed the study prior to phase II.
Arm/Group | Phase I Dose Level 1: 1200mg Eligible Higher Risk (HR) Myelodysplastic Syndromes (MDS) Participants
Number analyzed (Participants) | 0

14. Secondary Outcome: Phase II: Leukemia Free Survival (LFS)
Description: LFS is defined as progression to acute myeloid leukemia (AML) or death from any cause using the Kaplan-Meier method. Progression was assessed by the 2006 International Working Group response criteria for Myelodysplastic Syndromes using the Kaplan-Meier method and is defined as less than 5% blasts: ≥50% increase in blasts to >5% blasts; 5%-10% blasts: ≥50% increase to 10% blasts; 10%-20% blasts: ≥50% increase to >20% blasts; 20%-30% blasts: ≥50% increase to >30% blasts and any of the following: At least 50% decrement from maximum remission/response in granulocytes or platelets, reduction in Hgb by ≥2 g/dL, and transfusion dependence.
Time Frame: Until study closure
Population: This outcome measure was not done because the company closed the study prior to phase II.
Arm/Group | Phase I Dose Level 1: 1200mg Eligible Higher Risk (HR) Myelodysplastic Syndromes (MDS) Participants
Number analyzed (Participants) | 0

15. Secondary Outcome: Phase II: Overall Survival (OS)
Description: OS is defined as death from any cause using the Kaplan-Meier method.
Time Frame: Until study closure
Population: This outcome measure was not done because the company closed the study prior to phase II.
Arm/Group | Phase I Dose Level 1: 1200mg Eligible Higher Risk (HR) Myelodysplastic Syndromes (MDS) Participants
Number analyzed (Participants) | 0

16. Other Pre Specified Outcome: Number of Participants With Serious and/or Non-serious Adverse Events Assessed by the Common Terminology Criteria for Adverse Events (CTCAE v5.0)
Description: Here is the number of participants with serious and/or non-serious adverse events assessed by the Common Terminology Criteria for Adverse Events (CTCAE v5.0). A non-serious adverse event is any untoward medical occurrence. A serious adverse event is an adverse event or suspected adverse reaction that results in death, a life-threatening adverse drug experience, hospitalization, disruption of the ability to conduct normal life functions, congenital anomaly/birth defect or important medical events that jeopardize the patient or subject and may require medical or surgical intervention to prevent one of the previous outcomes mentioned.
Time Frame: From first study intervention, study day 1, through study day 100 after the end of the treatment cycle; approximately 7 months.
Population: 1/2 participants were enrolled but not treated.
Measure: Count of Participants; unit: Participants
Arm/Group | Phase I Dose Level 1: 1200mg Eligible Higher Risk (HR) Myelodysplastic Syndromes (MDS) Participants
Number analyzed (Participants) | 1
Participants | 1

17. Other Pre Specified Outcome: Phase I: Proportion of Participants With Dose-limiting Toxicities (DLT)
Description: DLT is defined as any of the following: ang grade ≥ non-hematologic toxicity that is possibly, probably, or definitely related to study drug. Liver injury as defined by a positive Hy's Law. And adverse reaction that leads to dose reduction or withdrawal.
Time Frame: First 28 days
Population: 1/2 participants were enrolled but not treated.
Measure: Number; unit: proportion of participants
Arm/Group | Phase I Dose Level 1: 1200mg Eligible Higher Risk (HR) Myelodysplastic Syndromes (MDS) Participants
Number analyzed (Participants) | 1
proportion of participants | 0

ADVERSE EVENTS:
Time Frame: From first study intervention, study day 1, through study day 100 after after the end of the treatment cycle; approximately 7 months.
Description: 1/2 participants were enrolled but not treated.
Arm/Group | Phase I Dose Level 1: 1200mg Eligible Higher Risk (HR) Myelodysplastic Syndromes (MDS) Participants
All-Cause Mortality (participants affected / at risk) | 0/1
Serious Adverse Events (participants affected / at risk) | 1/1
Other Adverse Events (participants affected / at risk) | 1/1
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase I Dose Level 1: 1200mg Eligible Higher Risk (HR) Myelodysplastic Syndromes (MDS) Participants (N=1)
Febrile neutropenia (Blood and lymphatic system disorders) | 1 (1)
Osteonecrosis of jaw (Musculoskeletal and connective tissue disorders) | 1 (1)
Skin infection (Infections and infestations) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Phase I Dose Level 1: 1200mg Eligible Higher Risk (HR) Myelodysplastic Syndromes (MDS) Participants (N=1)
Lymphocyte count decreased (Investigations) | 1 (1)
Neutrophil count decreased (Investigations) | 1 (1)
White blood cell decreased (Investigations) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol and Statistical Analysis Plan (2025-08-08): https://cdn.clinicaltrials.gov/large-docs/34/NCT05148234/Prot_SAP_004.pdf
  • Informed Consent Form: Cohort Screening Consent (2023-04-18): https://cdn.clinicaltrials.gov/large-docs/34/NCT05148234/ICF_001.pdf
  • Informed Consent Form: Cohort Affected Patient, Treatment (2023-12-21): https://cdn.clinicaltrials.gov/large-docs/34/NCT05148234/ICF_005.pdf